CLINICAL TRIAL: NCT04904666
Title: Safety and Efficacy of Bleach Baths in Non Critical Hospitalized Patients
Status: Completed | Type: Observational
Sponsor: Hospital Universitario Dr. Jose E. Gonzalez (Other)
Responsible Party: Principal Investigator, Dr. Adrian Camacho-Ortiz, Head of Infectious Diseases Department, Hospital Universitario Dr. Jose E. Gonzalez
Other Study IDs: IF19-00010
Record Dates: First submitted 2021-02-22; First posted 2021-05-27 (Actual); Last update posted 2021-05-27 (Actual); Status verified 2021-05

CONDITIONS: Safety Issues

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Bleach baths with .0125%
- Clorhexidine 2%
- Soap and water
- Bleach baths with .005%

SUMMARY:
Non critical hospitalized patients were bathed daily with 4 substances: bleach at .005%, bleach at .0125%, clorhexidine 2% and soap and water.

76 patients were enrolled and divided 19 subjects per group. Each patient was cultured with swab technique in palm, antecubital fold and armpit at day 0, day 3 and day 7 of enrollment.

Bacterial cultures were incubated and compared if decolonization occurred. Adverse events were evaluated in all patients.

Only 1 patient had and adverse event and was dry skin. Before patient was enrolled, he had dry skin because of his baseline disease. Moisturizing lotion was applied and patient continue in the study.

ELIGIBILITY:
Inclusion Criteria:

* Non critical hospitalized patients in internal medicine
* 18 years old and older

Exclusion Criteria:

* Burn patients
* Pregnant women
* Chloride hypersensitivity

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Non critical hospitalized patients in internal medicine that met inclusion criteria. Subjects should be hospitalized por 1 week.
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2019-11-26 (Actual); Primary Completion 2020-10-26 (Actual); Study Completion 2020-10-26 (Actual)

PRIMARY OUTCOMES:
Safety of Bleach baths as determined by the incidence of adverse or serious adverse events | November 26, 2019 - October 25, 2020

SECONDARY OUTCOMES:
Identification of bacterial colonization from pathogens belonging to the ESKAPE group | November 26, 2019 - October 25, 2020
  Identification of colonization by Enterococcus faecium, Staphylococcus aureus, Klebsiella pneumoniae, Acinetobacter baumannii, Pseudomonas aeruginosa and Enterobacter species
Percentage of patients remaining colonized 3, 5 and 7 days after daily baths | November 26, 2019 - October 25, 2020

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario José E. Gonzalez, Monterrey, Nuevo León, Mexico

IPD SHARING:
Plan to Share IPD: No